CLINICAL TRIAL: NCT00652808
Title: Double-Blind, Double Dummy, Randomized Comparison Study to Evaluate the Efficacy and Safety of Valdecoxib 10 mg QD and Naproxen 500 mg BID in Treating the Signs and Symptoms of Osteoarthritis of the Knee
Brief Title: Double-Blind, Double Dummy, Randomized Comparison Study to Evaluate the Efficacy and Safety of Valdecoxib 10 mg Once Daily and Naproxen 500 mg Twice Daily in Treating the Signs and Symptoms of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3471045
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis; Knee
Keywords: knee, OA patients
MeSH Terms: conditions — Osteoarthritis | interventions — valdecoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: naproxen

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 10 mg tablet by mouth once daily for 6 weeks
  Arms: Arm 1
Drug: naproxen — naproxen 500 mg capsule by mouth twice daily for 6 weeks
  Arms: Arm 2

SUMMARY:
This study was performed to demonstrate that treatment with valdecoxib 10 mg daily (QD) was at least as effective as with naproxen 500 mg twice daily (BID), a standard non-steroidal anti-inflammatory drug (NSAID), when taken for 6 weeks in Korean subjects with symptomatic osteoarthritis (OA) of the knee. Secondary objectives were to assess the overall safety and tolerability of valdecoxib 10 mg QD taken for 6 weeks in Korean subjects with symptomatic OA of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Korean outpatients with symptomatic radiologic evidence of OA of the knee (diagnosed according to the modified American College Rheumatology criteria)
* Patient's Assessment of Arthritis Pain measurement of at least 40 mm on VAS
* Patients had not received any NSAIDs or analgesics within 2 days (within 4 days for subjects taking oxaprozin, piroxicam or full dose aspirin) prior to the Baseline Visit

Exclusion Criteria:

* Diagnosis of inflammatory arthritis, gout, pseudogout, Paget's disease, or any chronic pain syndrome that, in the Investigator's opinion, would interfere with the assessment of the Index Knee
* Symptomatic anserine bursitis or acute joint trauma of the Index Knee
* Arthroscopy performed on the Index Knee within the past 12 months
* Complete loss of articular cartilage of the Index Knee
* Administration of oral, or intramuscular, intravenous, or soft tissue injections of corticosterosteroids within 4 weeks prior to screening visit
* Administration of intra-articular injection of corticosteroids or hyaluronic acid preparation in the Index Knee within 3 months or 6 months, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2004-05; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Patient's Assessment of Arthritis Pain using a Visual Analogue Scale (OA-Pain VAS) | Week 6

SECONDARY OUTCOMES:
WOMAC OA Physical Function | Week 2 and Week 6
WOMAC OA Stiffness Index | Week 2 and Week 6
Patient's Assessment of Arthritis Pain using a Visual Analogue Scale (OA-Pain VAS) | Week 2
Patient's Global Assessment of Arthritis Pain using a Visual Analogue Scale (OA-Pain VAS) | Week 2 and Week 6
adverse events | Continuous
Physician's Global Assessment of Arthritis Pain | Week 2 and Week 6
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) Osteoarthritis (OA) Composite Index | Week 2 and Week 6
WOMAC OA Pain Index | Week 2 and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- South Korea (5):
  - Pfizer Investigational Site, Anyang
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Pusan
  - Pfizer Investigational Site, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3471045&StudyName=Double-blind%2C%20double%20dummy%2C%20randomized%20comparison%20study%20to%20evaluate%20the%20efficacy%20and%20safety%20of%20Valdecoxib%2010%20mg%20once%20daily%20and%20Napro